CLINICAL TRIAL: NCT07105774
Title: The Effects of Stress Inoculation Training Program on Occupational Stress Level, Coping Style, and Sleep Quality in New Psychiatric Nurses：A Randomized Controlled Trial.
Brief Title: The Effects of Stress Inoculation Training Program on Occupational Stress Level, Coping Style, and Sleep Quality in New Psychiatric Nurses.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Huzhou University (Other)
Responsible Party: Principal Investigator, TianLe Xiang, Senior Nurse, Huzhou University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 202401-37
Record Dates: First submitted 2025-07-27; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Nurse; Psychiatric; Stress Inoculation Training

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The control group received routine training (Placebo Comparator): routine theoretical knowledge training and clinical practice training.
  Interventions: Behavioral: routine training
- The intervention group received the SIT program (Experimental): Establishment of online training groups, Establishment of stress reduction workshops and peer support groups, Organization of recreational activities and games for groups, ntroducing the concept, the program's curriculum, and process organization, Cognitive restructuring training, Relaxation training, Setting up virtual stressful situations and conducting stress resilience exercises, Self-reinforcement and consolidation, Applying competencies to solve practical problems, Recall and consolidation of course content
  Interventions: Behavioral: stress inoculation training program

INTERVENTIONS:
Behavioral: stress inoculation training program — The intervention group received the SIT program for 12 weeks. From 1st-2nd weeks, participants were admitted to an online training group set up via DingTalk, attending an offline stress reduction workshop were grouped into groups of 5-6, with games and small activities to promote group bonding. Psychiatric-psychological nurse specialist introduced the participants to the concept of SIT, the curriculum, and asked them to describe their initial knowledge and understanding of SIT. In addition, through cognitive restructuring training, the participants were made to review their work experience, understand the work stress and psychological pain they faced, and correctly recognize the role of cognition and emotion in causing and maintaining stress. From 3rd-6th weeks, participants were portrayed and discussed through videos and images, exploring personal, organizational and environmental stressors for new psychiatric nurses. Psychiatrists led relaxation exercises (e.g. positive thinking, med
  Other Names: stress inoculation training
  Arms: The intervention group received the SIT program
Behavioral: routine training — The control group received training in accordance with the "New Entry Nurse Training Syllabus (Trial)", which included routine theoretical knowledge training and clinical practice training.
  Arms: The control group received routine training

SUMMARY:
The aim of this clinical trial is to find out whether a stress inoculation program can reduce occupational stress in new psychiatric nurses. The main question it aimed to answer was:

Does a stress inoculation training program improve participants' occupational stress, coping styles, and sleep quality? The researchers compared the stress inoculation training to a conventional training control to see if the stress inoculation training reduced occupational stress.

ELIGIBILITY:
Inclusion Criteria:

* obtained nurse practitioner's license;
* nurses who were newly employed within the last three years and have been in their position for one month or longer;
* directly interacting with patients with mental illnesses in daily work;
* obtained informed consent to participate voluntarily in this study.

Exclusion Criteria:

* non-fresh graduates;
* these taking vacations, refresher courses during the study period;
* were breastfeeding or pregnant;
* had attended a similar stress intervention training (e.g., Positive Thinking Stress Reduction training, etc.) within the past year;
* new major non-work stressors (e.g., death of a close family member, divorce, exposure to a major natural disaster, etc.) within the last six months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2024-09-07 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-02-03 (Actual)

PRIMARY OUTCOMES:
Job stress scale for newly-graduated nurses (JSSNGN) | From enrollment to the end of treatment at 12 weeks
  Job stress scale for newly-graduated nurses (JSSNGN) is used to measure the level of occupational stress among new nurses. The scale consists of 4 dimensions and 24 items, including tasks in general care (9 items), tasks in critical care (4 items), interpersonal relationships (5 items), and leadership and management (6 items), and is based on a Likert's 5-point scale, ranging from "not stressful at all" to "extremely stressful", with Cronbach's α=0.93. JSSNGN was used to measure the level of occupational stress of new psychiatric nurses in this study. The scale has a total score range of 24 to 120, with higher scores representing greater occupational stress.

SECONDARY OUTCOMES:
Simplified Coping Style Questionnaire (SCSQ) | From enrollment to the end of treatment at 12 weeks
  Simplified coping style questionnaire (SCSQ) is designed to measure an individual's coping style in the face of a stressful event. Two subscales are active coping (problem-focused, SCSQ-A) and passive coping (emotion-focused, SCSQ-P) with items 1to12 for active coping strategies (problem-focused, SCSQ-A) and items 13 to 20 for passive coping strategies (emotion-focused, SCSQ-P). Each item uses a 4-point Likert's scale ranging from 0 to 3, from "not used" to "use frequently", with Cronbach's α=0.80 and correlations of test-retest reliability of 0.89. SCSQ was used to measure the coping styles (SCSQ-A and SCSQ-P respectively) of new psychiatric nurses when faced with occupational stress in this study, with higher scores indicating more frequent use of the coping style.
Pittsburgh sleep quality index (PSQI) | From enrollment to the end of treatment at 12 weeks
  Pittsburgh sleep quality index (PSQI) is used to measure the quality of an individual's sleep in the last 1 month. The scale consists of 19 self-assessed and 5 other-assessed items, of which the 19th self-assessed and 5 other-assessed items are not involved in scoring. The 18 self-assessed entries involved in scoring can be categorized into 7 dimensions: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction, each of which is scored on a 4-point scale from 0 to 3, and the cumulative score for each dimension is the total PSQI score, with a Cronbach's α = 0.85. PSQI was used to measure the sleep quality of the new psychiatric nurses in this study, with a total score of 0 to 21 points, with higher scores representing poorer sleep quality.

CONTACTS AND LOCATIONS:
Locations (1):
- Huzhou University, Huzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes